CLINICAL TRIAL: NCT02454166
Title: The Study of Chinese Medical Syndromes on Common Diseases: The Analysis of Chinese Medical Syndromes Differentiation on Acute Ischemic Stroke
Brief Title: The Analysis of Chinese Medical Syndromes Differentiation on Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 104-2081B
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ischemic stroke TCM syndromes Diagnostic Scale — A scale for Chinese medical differentiation
Other: Meridian Energy Analysis Device — A Device to assess involving meridian in certain diseases

SUMMARY:
Background and objective: Stroke, which means sudden onset of cerebral vascular accident. The earliest document was found in "Neijing". The ancient physicians had different opinions and points of view on the etiology and pathogenesis of stroke. Before the Tang and Song dynasty, the "exopathic wind" theory was talked about. And, after then, the "endogenous wind" theory was put forward. While in the Ming dynasty, Zhang Jing-Yue advocated that "Stroke is not caused by wind etiology'', highlighting the much difference of the thinking. Until nowadays, many famous physicians have their own unique way to determine the etiologic factor based on differentiation. To be practical, objectivity differentiating and determining the etiologic factor of stroke is the foundation of establishing the treatment guidelines. The investigators aim to establish the scientific epidemiological standard of traditional Chinese Medicine (TCM) syndromes of acute ischemic stroke in Taiwan.

DETAILED DESCRIPTION:
Methods: The investigators use the ischemic stroke TCM syndromes Diagnostic Scale (ISTCMDS) and the Meridian Energy Analysis Device (M.E.A.D.) to objectively analyze the diagnostic elements and detect the deficiency or excess performance of meridians of acute ischemic stroke patients from Stroke Center at Linkou Chang Gung Memorial Hospital. The onset of stroke is set Within 7 days, and the investigators expected to collect 300 patients. The investigators initially establish the scientific epidemiological study of acute ischemic stroke with TCM syndromes and deficiency or excess of meridian performances through statistical analysis to become a standard of Chinese and Western medicine integration. The data collection can gradually become a library, which will facilitate the assessment of the clinical efficacy of TCM adjuvant therapy and become a basis to assist Western and Chinese medicine integration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute ischemic stroke, approved by brain CT or MRI
* Onset within 7 days
* No other severe organic diseases
* Stroke for the first time or recurrent stroke with previous Rankin's scale ≦1 status
* Signed Inform Consent

Exclusion Criteria:

* Not meet the above diagnostic and inclusion criteria
* Complicated with sepsis or other infections
* Refuse to accept Chinese Medical syndromes differentiation, the Meridian Energy Analysis Device (M.E.A.D.), or refuse to sign Inform Consent
* Unconsciousness
* With pacemaker or pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute ischemic stroke patients from Stroke Center at Linkou Chang Gung Memorial Hospital. The onset of stroke is set Within 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Chinese medical syndromes differentiation by Ischemic stroke TCM syndromes Diagnostic Scale (ISTCMDS) in acute stroke patients | within 7 days from the onset of the stroke

CONTACTS AND LOCATIONS:
Overall Officials: Shu-chen Cheng, Study Chair — Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital at Linkou; YEU-JHY CHANG, Study Chair — Stroke Center and Department of Neurology, Chang Gung Memorial Hospital at Linkou